CLINICAL TRIAL: NCT07154368
Title: A Randomized, Open-Label, Multicenter, Phase 3 Study Evaluating the Efficacy and Safety of JYP0322 Versus Platinum-Based Chemotherapy in ROS1-Positive Locally Advanced or Metastatic Non-Small Cell Lung Cancer Patients Previously Treated With ROS1-TKI Therapy.
Brief Title: JYP0322 Versus Platinum Based Doublet Chemotherapy in ROS1 Positive Patients Previously Treated With ROS1-TKIs.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guangzhou JOYO Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JYP0322M302
Record Dates: First submitted 2025-08-19; First posted 2025-09-04 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Pemetrexed

STUDY DESIGN:
Intervention Model Description: two arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JYP0322 tablets (Experimental)
  Interventions: Drug: JYP0322 tablets
- Pemetrexed Disodium (Experimental)
  Interventions: Drug: Pemetrexed injection; Drug: Cross-over to JYP0322

INTERVENTIONS:
Drug: Pemetrexed injection — Randomization to either JYP0322 or platinum-based doublet-chemotherapy on Day 1 of every 21d cycle in a 2:1 (JYP0322: platinum-based doublet-chemotherapy) ratio
  Arms: Pemetrexed Disodium
Drug: Cross-over to JYP0322 — Once subjects on the platinum-based doublet chemotherapy arm are determined to have objective radiological progression according to RECIST 1.1 by the investigator and confirmed by BICR, they will be given the opportunity to begin treatment with JYP0322 150mg tid. These subjects may continue treatment with JYP0322 if they are continuing to show clinical benefit until disease progression as judged by the investigator.
  Arms: Pemetrexed Disodium
Drug: JYP0322 tablets — JYP0322, 150 mg, administered orally three times daily (tid) after meals; sample size (N) = 60.
  Arms: JYP0322 tablets

SUMMARY:
The primary purpose of the study was to compare progression-free survival of JYP0322 vs. platinum-based doublet chemotherapy in patients previously treated with ROS1-TKIs. Patients in the chemotherapy arm are given the option to switch to JYP0322 after BICR confirmed progressive disease (PD), while also have the choice to pursue with other drugs after discussing with their physicians.

DETAILED DESCRIPTION:
This is a phase III, open label, randomized study assessing JYP0322 (150 mg, orally, tid) versus platinum-based doublet chemotherapy in subjects with confirmed diagnosis of ROS1 fusion positive NSCLC, who have progressed following prior therapy with one or two approved ROS1 Tyrosine Kinase Inhibitor (ROS1-TKI) agents and whose tumors harbors a ROS1 fusion positive. Subjects must agree to provide a biopsy for central confirmation of ROS1 fusion status. A total of 207 patients will be randomly assigned in a 2:1 ratio to receive oral JYP0322 (at a dose of 150mg tid) or intravenous pemetrexed (500 mg per square meter of body-surface area) plus carboplatin (target area under the curve 5 [AUC5]) every 3 weeks for up to six cycles. Patients without disease progression after four cycles of platinu

ELIGIBILITY:
Inclusion Criteria:

* Key Inclusion Criteria

  * Subjects with histologically or cytologically documented NSCLC.
  * Locally advanced or metastatic ROS1 fusion positive NSCLC.
  * Prior one or two ROS1-TKI(s) Treatment.
  * World Health Organization (WHO) performance status 0-1.
  * Life expectancy of at least 3 months.
  * At least one measurable lesion according to RECISIT 1.1.

Exclusion Criteria:

* Key Exclusion Criteria:

  * Current participation in another therapeutic clinical trial.
  * Gastrointestinal disease (e.g., Crohn's disease, ulcerative colitis, or short gut syndrome) or other malabsorption syndromes that would impact on drug absorption.
  * A history of severe allergies, or a history of severe allergy, hypersensitivity or other hypersensitivity to any active or inactive ingredient of the study drug.
  * All acute toxic effects (excluding alopecia) of any prior anti-cancer therapy to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0 Grade more than 1.
  * Any investigational agents or other anticancer drugs from a previous treatment regimen or clinical study within 14 days of the first dose of study treatment.
  * Known active infe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2025-09-23 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) by BICR Assessment | UP to 3 years
  Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Progressive Disease (PD): >= 20% increase in the sum of diameters of TLs and an absolute increase in sum of diameters of >=5mm (compared to the previous minimum sum) or progression of NTLs or a new lesion. PFS is the time from date of randomization until the date of PD (by BICR assessment) or death (due to any cause) regardless of whether the patient withdrew from randomized therapy. Patients who had not progressed or died at the time of analysis were censored at the time of the latest date of assessment from their last evaluable RECIST 1.1 assessment.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) by investigators Assessment | UP to 3 years
  Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) assessed by MRI or CT: Progressive Disease (PD): >= 20% increase in the sum of diameters of TLs and an absolute increase in sum of diameters of >=5mm (compared to the previous minimum sum) or progression of NTLs or a new lesion. PFS is the time from date of randomization until the date of PD (by investigators assessment) or death (due to any cause) regardless of whether the patient withdrew from randomized therapy. Patients who had not progressed or died at the time of analysis were censored at the time of the latest date of assessment from their last evaluable RECIST 1.1 assessment
Overall Survival (OS) | UP to 5 years
  OS is defined as the time from date of randomization until the date of death (due to any cause) regardless of whether the patient withdrew from randomized therapy. Patients who had not died would be censored at the last known alive date.
Objective Response Rate (ORR) by Investigator and BICR assessment | RECIST tumor assessments every 6 weeks from randomization up to 3 years.
  Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions. ORR is the percentage of patients with at least 1 visit response of CR or PR prior to progression or any further therapy.
Duration of Response (DOR) by Investigator and BICR assessment | RECIST tumor assessments every 6 weeks from randomization up to 3 years.
  Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions. DOR is the time from the date of first documented response until the date of documented progression or death in the absence of disease progression for patients who had conformed CR or PR.
Disease Control Rate (DCR) by Investigator and BICR assessment | RECIST tumor assessments every 6 weeks from randomization up to 3 years.
  Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions; Stable disease (SD): Neither sufficient shrinkage to qualify as a response nor sufficient growth to qualify as progression; Progressive Disease (PD): >= 20% increase in the sum of diameters of TLs and an absolute increase in sum of diameters of >=5mm (compared to the previous minimum sum) or progression of NTLs or a new lesion. DCR is the percentage of patients with best response of CR, PR or SD at >=6 weeks, prior to any progressive disease (PD).
Time to Response (TTR) by Investigator and BICR assessment | RECIST tumor assessments every 6 weeks from randomization up to 3 years.
  Per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions; Stable disease (SD): Neither sufficient shrinkage to qualify as a response nor sufficient growth to qualify as progression; TTR is defined as time from the date of randomization to the first documented response for patients who had confirmed CR or PR at least once.

IPD SHARING:
Plan to Share IPD: No